CLINICAL TRIAL: NCT03452813
Title: Transitions of Care Stroke Disparity Study (TCSD-S)
Acronym: TCSD-S
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Jose Romano, MD, Principal Investigator, University of Miami
Other Study IDs: 20170892; 1R01MD012467 (NIH); 20170892 (Other: IRB)
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Stroke
Keywords: transitions of care; stroke disparities
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ischemic stroke or intracerebral hemorrhage patients: patients discharged from hospital to home or discharged to rehab will be called at 30 day and 90 day to monitor their transition of care outcomes.

SUMMARY:
The TCSD Study will identify disparities in transitions of stroke care and key factors associated with effective transitions of care through structured telephone interviews to evaluate medication adherence, healthy lifestyle, utilization of rehabilitation interventions and medical follow-up 30 days after hospital discharge to home in 2,400 participants across 12 comprehensive stroke centers (CSC) in Florida. A novel Transitions of Stroke Care Performance Index (TOSC PI) correlated with 90-day rehospitalization will be derived and validated.

DETAILED DESCRIPTION:
The TCSD Study will identify disparities in transitions of stroke care and key factors associated with effective transitions of care through structured telephone interviews to evaluate medication adherence, healthy lifestyle, utilization of rehabilitation interventions and medical follow-up 30 days after hospital discharge to home and in-patient care rehabilitation in 2,400 participants across 12 comprehensive stroke centers (CSC) in Florida. A novel Transitions of Stroke Care Performance Index (TOSC PI) will be derived and validated. The primary outcomes are the TOSC PI and 90-day readmission. Other stroke outcomes include stroke disability, recurrence, cardiovascular events, and death at 3 months. Outcomes will be collected through telephone interviews and review of patient charts. Predictors of disparities in transition of care and outcomes will be evaluated using baseline in-hospital data during acute stroke hospitalization obtained from the Florida Stroke Registry and Social Determinants of Health obtained through novel data collected from publicly available records. Based on identified predictors of disparities in TOSC, we will develop and demonstrate feasibility of initiatives for interventions to reduce disparities in TOSC that target systems of care with a TOSC disparities dashboard, and health care providers with a training module for enhanced education and support at discharge and during follow-up. We will evaluate any temporal improvements in the TOSC Performance Index and outcomes before and after the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke or intracerebral hemorrhage patients age >/=18 years that are discharged directly to home, or discharged to rehab
* Final diagnosis of ischemic stroke or intracerebral hemorrhage, included in the Get With
* The Guidelines- Stroke (GWTG-S) database.
* Patient or legally authorized representative provides consent
* Available by phone and willing to receive two follow-up calls.

Exclusion Criteria:

* Cases with subarachnoid hemorrhage, transient ischemic attack (TIA), stroke not otherwise specified, no stroke related diagnosis, and admission for elective carotid intervention will be excluded.
* Prisoners will be excluded. The purpose of the project is to study the hospital-to-home transition of stroke care.
* Discharged to inpatient rehabilitation, nursing home, subacute rehabilitation facilities or assisted living facilities. These facilities support medication adherence, provide prescribed diets, often provide in-house medical follow-up, and therefore disparities in TOSC are less likely to be detected and not amenable to the proposed interventions.
* Modified Rankin Scale of 0 after stroke. These individuals usually do not require any rehabilitation interventions and to avid the inclusion of predominately mild stroke patients.
* Unable to obtain consent from patient or legally authorized representative.
* Unavailable or unwilling to participate in the 30 and 90 day follow up telephone calls.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The TCSD-S participating study sites (SS) include 6 Comprehensive Stroke Centers (CSC) that currently participate in the Florida Stroke Registry will be Study. The SS will identify and consent participants and collect TOSC performance metrics and outcomes. A total of 2,400 ischemic stroke and intracerebral hemorrhage participants from 6 Florida CSC that are discharged directly to home will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1549 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Transitions of Stroke Care Performance Index | 30 days
  Transitions of Stroke Care Performance Index (TOSC-PI) is a novel score that will be developed based on the results of this study to predict effective transitions of care, and will be composite score that includes medication and lifestyle adherence, diet, tobacco and alcohol cessation, exercise, utilization of rehabilitation services, and medical follow-up after discharge. The index will be calculated as the points achieved over the total for which the participant is eligible. High scores indicate successful transition of care, while low scores reflect inadequacies and gaps in transitions of care.
Hospital readmission | 90 days
  Review and documentation of the participants readmission to hospital within 90 days post discharge

SECONDARY OUTCOMES:
Modified Rankin Scale (mRS) | 90 days
  Measurement of participants degree of disability/dependence in daily activities. The scale runs from 0 (No symptoms at all) to 6 (dead).
Stroke recurrence | 90 days
  documentation of the number of times a participant has experienced another stroke.
Cardiovascular events | 90 days
  incident cardiovascular events
Mortality rate | 90 days
  number of deaths

CONTACTS AND LOCATIONS:
Overall Officials: Jose G Romano, MD, Principal Investigator — UNIVERISTY OF MIAMI
Locations (2):
- United States (2):
  - Jackson Memorial Hospital, Miami, Florida
  - University of Miami, Miami, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dong C, Gardener H, Rundek T, Marulanda E, Gutierrez CM, Campo-Bustillo I, Gordon Perue G, Johnson KH, Sacco RL, Romano JG; Transitions of Care Stroke Disparities Study (TCSD-S) Investigatorsdagger. Factors and Behaviors Related to Successful Transition of Care After Hospitalization for Ischemic Stroke. Stroke. 2023 Feb;54(2):468-475. doi: 10.1161/STROKEAHA.122.040891. Epub 2022 Dec 19. PMID 36533520